CLINICAL TRIAL: NCT01657734
Title: Multimodal MR Imaging in Patients With Glioblastoma Treated With Dendritic Cell Therapy
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S53303
Record Dates: First submitted 2011-09-07; First posted 2012-08-06 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Malignant Gliomas
Keywords: therapy-induced inflammatory response with; magnetic resonance imaging
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- HGG2003: **** patients enrolled in the HGG 2003 HGG-IMMUNO 2003 trial
  Patients, older than 3 and younger than 60 years with relapse of high-grade glioma (anaplastic astrocytoma WHO grade III or glioblastoma multiforme WHO grade IV), histologically diagnosed in the first stage of the disease as well as after relapse or relapse of glioma which was grade II in the First phase but grade III or IV upon relapse are treated with dendritic cell therapy (immunotherapy) as single treatment approach (No radiotherapy and/or chemotherapy).
  Interventions: Other: MR imaging
- HGG2010: **** patients enrolled in the HGG 2010 HGG-IMMUNO 2010 trial
  * prospective double blind placebo controlled randomised clinical trial HGG-2010 for patients with newly diagnosed glioblastoma in which immunotherapy is integrated in the current standard of care (concommitant radiochemotherapy).
  Interventions: Other: MR imaging

INTERVENTIONS:
Other: MR imaging — MR imaging

SUMMARY:
Malignant gliomas are aggressive tumours with poor prognosis despite the current multimodal treatment. Hence, there is a clear need for new, effective therapies, among which immune therapy has emerged as a promising treatment option.

When interpreting follow-up magnetic resonance (MR) examinations, the radiologist is often confronted with images that are difficult to interpret with the conventional anatomical imaging techniques. The difference between tumour relapse and therapy-mediated changes is not always distinctive.

In this project, the investigators attempt to characterize the inflammatory response with parameters from advanced MRI techniques like MR spectroscopy, MR perfusion imaging and MR-diffusion imaging. These techniques allow characterization of cellular properties like metabolism and tissue structure respectively. Doing so, the investigators will monitor disease evolution in order to timely detect treatment failure, thereby allowing appropriate switch in patient management.

ELIGIBILITY:
Inclusion Criteria:

**** patients enrolled in the HGG 2003 HGG-IMMUNO 2003 trial

Patients, older than 3 and younger than 60 years with relapse of high-grade glioma (anaplastic astrocytoma WHO grade III or glioblastoma multiforme WHO grade IV), histologically diagnosed in the first stage of the disease as well as after relapse or relapse of glioma which was grade II in the First phase but grade III or IV upon relapse are treated with dendritic cell therapy (immunotherapy) as single treatment approach (No radiotherapy and/or chemotherapy).

**** patients enrolled in the HGG 2010 HGG-IMMUNO 2010 trial

* prospective double blind placebo controlled randomised clinical trial HGG-2010 for patients with newly diagnosed glioblastoma in which immunotherapy is integrated in the current standard of care (concommitant radiochemotherapy).

Exclusion Criteria:

minor age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with glioblastoma treated with dendritic cell therapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-02-18 (Actual); Study Completion 2016-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - University Hospitals Leuven, Leuven, Vlaams-Brabant
  - University Hospitals of Leuven, Leuven, Vlaams-Brabant